CLINICAL TRIAL: NCT00727870
Title: A Single Site, Three Arm, Open Label Comparative Preference Study to Evaluate the Preference of Consumers and Health Care Professionals for the Use of Shapes by PolyMem Wound Dressings and Shapes by PolyMem Silver Wound Dressings, Each Compared to Antibiotic Ointment Covered With a Band-aid Type Dressing (Current Standard of Practice) and to Each Other in the Post-biopsy Management of Shave Biopsies. Each Participant Serves as Own Control. A Blinded Third Party Physician Will Evaluate and Compare the Wounds Based on Photos Taken at the Various Follow-up Points..
Brief Title: Evaluation of Preferences of Consumers and Clinicians for the Management of Shave Biopsy Sites With a PolyMem Formulation Dressing or Current Standard of Care.
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ferris Mfg. Corp. (Industry)
Collaborators: Chicago Skin Clinic (Other); University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PolyMem001
Record Dates: First submitted 2008-07-31; First posted 2008-08-04 (Estimated); Last update posted 2012-03-02 (Estimated); Status verified 2012-03

CONDITIONS: Healing
Keywords: Shave Biopsy management; "Biopsy/adverse effects"[Mesh]; "Biopsy/complications"[Mesh])

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Other): After the two biopsies, one site will be covered with the antibiotic ointment and the band-aid type bandage (physician's current standard of care) and the other site will be covered the Shapes by PolyMem dressing.
  Interventions: Device: Shapes by PolyMem dressing
- 2 (Other): Arm 2: after the two biopsies, one site will be covered with the antibiotic ointment and the band-aid type bandage (physician's current standard of care) and the other site will be covered the Shapes by PolyMem Silver dressing.
  Interventions: Device: Shapes by PolyMem Silver Dressing
- 3 (Other): Arm 3: after the two biopsies, one site will be covered with Shapes by PolyMem dressing and the other site will be covered the Shapes by PolyMem Silver dressing.
  Interventions: Device: Shapes by PolyMem on one site and Shapes by PolyMem Silver dressing on second site

INTERVENTIONS:
Device: Shapes by PolyMem dressing — Shapes by PolyMem dressing on one site compared to antibiotic ointment covered with band-aid type dressing on second site
  Arms: 1
Device: Shapes by PolyMem Silver Dressing — Shapes by PolyMem Silver dressing on one site compared to antibiotic ointment covered with band-aid type dressing on second site
  Arms: 2
Device: Shapes by PolyMem on one site and Shapes by PolyMem Silver dressing on second site — Shapes by PolyMem dressing on one site. Shapes by PolyMem Silver dressing on other site.
  Arms: 3

SUMMARY:
Shave biopsies are often uncomfortable during the healing process. This is a preliminary study to determine if patients and clinicians prefer using PolyMem formulating dressings on shave biopsy sites compared to the current standard of practice, which is antibiotic ointment covered with a band-aid type dressing.

DETAILED DESCRIPTION:
Only individuals who require 2 shave biopsies on the same treatment day will be entered in the study. Each participant serves as their own control.

ELIGIBILITY:
Inclusion Criteria:

* Individuals that are going to have two shave biopsies performed on the same day will be evaluated for inclusion in the study.

Exclusion Criteria:

* Those that have used systemic corticosteroids in the last three months.
* Those with any medical condition leading to immunosuppression
* Those with a history of keloid formation
* Those with documented compromised wound healing potential
* History of psoriasis or eczema in the last 2 years
* Those with an active infection
* Those that use aspirin or non-steroidal anti-inflammatory drugs more than 3 times per week for pain (daily low dose aspirin use for cardiovascular health is not an exclusion criteria)
* Those that have inflammatory conditions such as rheumatoid arthritis or Crohn's disease
* Those that have clinical signs of malnutrition that could interfere with wound healing
* Those that have a history of allergies to any wound dressing or medical tape
* Those that are not able to change the dressing themselves and do not have anyone in their household that can change the dressings if needed.
* Those younger than 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2008-07; Primary Completion 2011-10 (Actual); Study Completion 2012-06 (Estimated)

PRIMARY OUTCOMES:
Preference by both clinician and consumer of dressing choice in managing shave biopsy sites. | At completion of protocol

SECONDARY OUTCOMES:
Evaluations and comparisons by both treating physician and blinded physician of each site for differences in inflammation, signs of possible infection, reepithelialization and cosmetic appearance | At completion of protocol

CONTACTS AND LOCATIONS:
Overall Officials: Andrew M Gorchynsky, MD, Principal Investigator — Chicago Skin Clinic; Danilo V Del Campo, MD, Principal Investigator — Chicago Skin Clinic
Locations (1):
- Chicago Skin Clinic, Chicago, Illinois, United States